CLINICAL TRIAL: NCT01110382
Title: A Prospective, Randomized, Double-Blind, Multicenter Study to Establish the Safety and Tolerability of Doripenem Compared With Meropenem in Hospitalized Children With Complicated Intra-Abdominal Infections
Brief Title: A Safety and Tolerability Study of Doripenem Compared With Meropenem in Children Hospitalized With Complicated Intra-abdominal Infections
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial terminated early per business decision
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016789; DORIPED3001 (Other: Janssen Research & Development, LLC); 2009-015864-32 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-04-15; First posted 2010-04-26 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Abscess, Intra-Abdominal; Abdominal Abscess; Abdomen, Acute; Abdominal Pain; Appendicitis; Rupture; Infection; Intestinal Perforation; Peritonitis; Ileus
Keywords: Anti-Infective Agents; Doripenem; Meropenem; Child, Hospitalized; Complicated Intra-Abdominal Infections
MeSH Terms: conditions — Abdominal Abscess; Abdomen, Acute; Abdominal Pain; Appendicitis; Rupture; Infections; Intestinal Perforation; Peritonitis; Ileus | interventions — Doripenem; Meropenem; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doripenem (Experimental): Doripenem 20 mg/kg per dose (up to 500 mg/dose)will be administered every 8 hours as 60-minutes IV (at least 3 days of IV doripenem only or IV doripenem followed by oral amoxicillin/clavulanate potassium). Total duration of treatment 5 to 14 days.
  Interventions: Drug: Doripenem; Drug: Meropenem placebo; Drug: Amoxicillin/clavulanate potassium
- Meropenem (Experimental): Meropenem 20 mg/kg per dose (up to 1 g/dose) will be administered every 8 hours as 30-minutes IV (at least 3 days of IV meropenem only or IV meropenem followed by oral amoxicillin/clavulanate potassium). Total duration of treatment 5 to 14 days.
  Interventions: Drug: Meropenem; Drug: Doripenem placebo; Drug: Amoxicillin/clavulanate potassium

INTERVENTIONS:
Drug: Doripenem — Type=once every 8 hours infused over 60 minutes, Unit=mg, Number=20mg/kg up to 500mg/dose, Form=solution for infusion, Route-intravenous use. At least 3 days of iv doripenem administered every 8 hours immediately after meropenem placebo for up to 14 days
  Arms: Doripenem
Drug: Meropenem placebo — Form=solution for infusion, Route=intravenous use, administered once every 8 hours infused over 30 minutes immediately before each iv infusion of doripenem for up to 14 days.
  Arms: Doripenem
Drug: Meropenem — Type=once every 8 hours infused over 30 minutes, Unit=mg, Number=20 mg/kg to 1 gram per dose, Form=solution for infusion, Route=intravenous use. At least 3 days of iv meropenem administered every 8 hours immediately before doripenem placebo for up to 14 days
  Arms: Meropenem
Drug: Doripenem placebo — Form=solution for infusion, Route=intravenous use, administered once every 8 hours infused over 60 minutes immediately after each iv infusion of meropenem for up to 14 days
  Arms: Meropenem
Drug: Amoxicillin/clavulanate potassium — Form=suspension or tablets, Route=oral (by mouth), may be administered at the discretion of the investigator once every 12 hours for up to 14 days following IV therapy with doripenem or meropenem.

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of doripenem compared with meropenem in children hospitalized with complicated intra-abdominal infections.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), double-blind (neither physician nor patient knows the name of the assigned study drugs), double-dummy (all patients are given both a placebo [salt solution] and study drug in alternating periods of time during the study), active comparator-controlled (compare the "test" treatment to standard-of-care therapy), multinational, multicenter study to evaluate the safety of the study drugs (doripenem and meropenem) administered by intravenous (iv) infusion (slow injection of drug solution into the vein over a period of time) in children aged 3 months to less than 18 years who are hospitalized with complicated intra abdominal infections (cIAI). Complicated intra abdominal infections include but are not limited to appendicitis with rupture and/or abscess (local collection of pus), acute (severe or intense) gastric, duodenal (beginning section of the small intestine), or gall bladder perforation (a hole in the wall of the stomach, small intestine, or gallbladder), and secondary peritonitis. The study will include 3 periods: a pretreatment (screening) period that will occur within 2 days prior to randomization (assignment of study drug), a treatment period of 5 to 14 days where patients will receive iv study drug treatment only or IV study therapy and a switch to oral antibiotic therapy, and a posttreatment period consisting of 2 study visits. The max duration of study drug therapy is 14 days. The total duration of the study is approximately 7 to 8 weeks. Safety and tolerability will be evaluated by examining the incidence, severity, and type of adverse events, changes in clinical laboratory tests, vital signs measurements, and findings from physical examinations observed during treatment and at each posttreatment visit. An independent monitoring committee (IDMC) will be established for this study to ensure that the safety of patients is not compromised. The IDMC will consist of individuals who are not associated with the conduct of the study, and will include but will not be limited to individuals with expertise relevant to the care of pediatric patients, and including at least one infectious disease physician and at least one statistician. Patients will receive IV Doripenem (20 mg/kg to 500 mg/dose) and meropenem placebo OR meropenem (20 mg/kg to 1 gram/dose) and doripenem placebo once every 8 hours for up to 14 days. If the patient's cIAI symptoms improve after 72 hours of treatment with iv study drug, the investigator may choose to stop iv study drug and switch the patient to an orally administered antibiotic (amoxicillin/clavulanate postassium) to complete the 5- to 14 day course of antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible for the study must have clinical evidence of cIAI
* Require surgical intervention (eg, laparotomy, laparoscopic surgery, or percutaneous drainage) to manage the cIAI
* Require antibacterial therapy for 5 to 14 days in addition to the surgical intervention
* Must, based on the judgment of the investigator, require hospitalization initially and antibacterial therapy for 5 to 14 days in addition to surgical intervention for the treatment of the current cIAI. (Note that the patient must require at least 3 days of IV antibiotic therapy initially)
* Have a signed informed consent form completed by the patient's parent or legal representative (and a signed assent form obtained from patients who are capable of providing assent, typically, children 7 years of age and older)

Exclusion Criteria:

* Have a history of hypersensitivity reactions to carbapenems, cephalosporins, penicillins, or other beta-lactam antibiotics
* concomitant infection including but not limited to suspected or confirmed meningitis or central nervous system infection requiring systemic antibiotic or antifungal therapy in addition to the iv study drug therapy at the time of randomization
* Receipt of nonstudy systemic antibiotic therapy for cIAI for more than 24 hours immediately preceding the start of the infusion of the first dose of iv study drug therapy
* Have a diagnosis of abdominal wall abscess confined to musculature of the abdominal wall, small bowel obstruction or ischemic bowel disease without perforation, traumatic bowel perforation requiring surgery within 12 hours of perforation, or perforation of gastroduodenal ulcers requiring surgery within 24 hours of perforation (these are considered situations of peritoneal soiling before the infection has become established)
* Have simple (noncomplicated), nonperforated appendicitis or gangrenous appendicitis without rupture into the peritoneal cavity identified during a surgical procedure OR presence of spontaneous bacterial peritonitis or peritonitis associated with cirrhosis or chronic ascites
* Known at the time of randomization to have a cIAI caused by at least one pathogen that is nonsusceptible to doripenem or meropenem
* Presence of any of the following clinically significant laboratory abnormalities: Hematocrit of less than 20%, absolute neutrophil count (ANC) <500 cells/µL, platelet count <40,000 cells/µL, serum alanine aminotransferase or aspartate aminotransferase (AST) or total bilirubin 5 times or greater the age-specific upper limit of normal (ULN) or acute/chronic renal insufficiency with a baseline creatinine clearance <50 mL per minute or requires dialysis therapy for any reason
* Have a history of uncontrolled epilepsy defined as at least 1 seizure within the 6 months before randomization

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2010-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (19):
- United States (4):
  - San Diego, California
  - Washington D.C., District of Columbia
  - Cleveland, Ohio
  - Toledo, Ohio
- Argentina (5):
  - Buenos Aires
  - Córdoba
  - Loma Hermosa
  - Paraná, Entre Ríos
  - Santa Fe
- Brazil (2):
  - Passo Fundo
  - São Paulo
- Chile (2):
  - Santiago
  - Valdivia X Región
- Colombia (2):
  - Bogotá
  - Floridablanca
- Riga, Latvia
- Lithuania (2):
  - Kaunas
  - Vilnius
- Zona, Panama

RESULTS

PARTICIPANT FLOW:
Groups:
- Doripenem: Doripenem 20 mg/kg per dose (up to 500 mg/dose) was administered every 8 hours as 60-minutes IV (at least 3 days of IV doripenem only or IV doripenem followed by oral amoxicillin/clavulanate potassium). Total duration of treatment 5 to 14 days.
- Meropenem: Meropenem 20 mg/kg per dose (up to 1 g/dose) was administered every 8 hours as 30-minutes IV (at least 3 days of IV meropenem only or IV meropenem followed by oral amoxicillin/clavulanate potassium). Total duration of treatment 5 to 14 days.
Period: Overall Study
Arm/Group | Doripenem | Meropenem
Started | 31 | 10
Completed | 31 | 8
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doripenem | Meropenem | Total
Number analyzed (Participants) | 31 | 10 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31 | 10 | 41
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.5 (3.40) | 9.3 (4.52) | 8.7 (3.66)
Age, Customized [Number; unit: participants]
  3 months to <2 years | 0 | 0 | 0
  2 to <6 years | 5 | 3 | 8
  6 to <12 years | 18 | 4 | 22
  12 to <18 years | 8 | 3 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 0 | 15
  Male | 16 | 10 | 26

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Clinical Cure Rate at Test Of Cure (TOC) Visit
Description: The participants were considered as clinical cure if they had clinical improvement in signs and symptoms of the intra-abdominal infection such that no additional antibacterial therapy or surgical or percutaneous intervention is/was required for the treatment of the index infection, no fever, and a favorable response at End of IV visit.
Time Frame: TOC (7 to 14 days after the last dose of study medication therapy)
Population: Clinical Intent-to-Treat (CITT): All randomized participants who met the minimal disease definition of complicated intra-abdominal infection regardless if a baseline pathogen was isolated from the intra-abdominal cavity.
Measure: Number; unit: participants
Arm/Group | Doripenem | Meropenem
Number analyzed (Participants) | 31 | 10
participants | 23 | 7

2. Secondary Outcome: The Number of Participants With Clinical Improvement Rate at End of IV (EIV) Visit
Description: The participants were considered as clinical improved if they had clinical improvement in signs and symptoms of the intra-abdominal infection, no fever, decrease in WBC, and not received any nonstudy antibiotics for the treatment of intra-abdominal infection after IV study drug therapy had begun.
Time Frame: EIV (within 24 hours after completion of the last dose of IV study medication therapy)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Doripenem | Meropenem
Number analyzed (Participants) | 31 | 10
participants | 29 | 8

3. Secondary Outcome: The Number of Participants With Clinical Cure Rate at Late Follow-Up (LFU) Visit
Description: as for outcome 1
Time Frame: LFU (28 to 42 days after the last dose of study medication therapy)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Doripenem | Meropenem
Number analyzed (Participants) | 31 | 10
participants | 22 | 6

4. Secondary Outcome: The Number of Participants With Favorable Per-participant Microbiological Response
Description: Favorable per-participant microbiological response rate was evaluated at the at End of IV (EIV) visit, Test Of Cure (TOC) visit, and Late Follow-Up (LFU) visit. The favorable per-participant microbiological response was considered when all baseline pathogens were eradicated (absence) or presumed eradicated (absence of material to culture in a participant who has a positive clinical response to treatment).
Time Frame: EIV (within 24 hours after completion of the last dose of IV study medication therapy), TOC (7 to 14 days after the last dose of study medication therapy), and LFU (28 to 42 days after the last dose of study medication therapy)
Population: Microbiological intent-to-treat - Participants of CITT with at least 1 baseline bacterial pathogen isolated from the intra-abdominal cavity that was susceptible to both doripenem and meropenem. 8 and 2 participants from doripenem and meropenem, respectively had no susceptible intra-abdominal pathogen at baseline and were excluded from this set.
Measure: Number; unit: participants
Arm/Group | Doripenem | Meropenem
Number analyzed (Participants) | 23 | 8
participants
  EIV visit | 21 | 6
  TOC visit | 17 | 5
  LFU visit | 17 | 5

5. Secondary Outcome: Number of Participants With Favorable Per-pathogen Microbiological Outcome Rate at End of IV (EIV) Visit
Description: A total of 24 pathogens in the doripenem group and 6 pathogens in the meropenem group were isolated at baseline from the intra-abdominal culture and were susceptible to the study drug received. The most common pathogens isolated from the intra-abdominal culture are listed in the table below; the numbers in parenthesis next to each pathogen represent the number of participants with the pathogen isolated at baseline in the doripenem and meropenem treatment groups, respectively. The favorable per-pathogen microbiological outcome was considered when all baseline pathogens were eradicated (absence) or presumed eradicated (absence of material to culture in a participant who has a positive clinical response to treatment).
Time Frame: EIV (within 24 hours after completion of the last dose of IV study medication therapy)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Doripenem | Meropenem
Number analyzed (Participants) | 23 | 8
participants
  Streptococcus anginosus (13, 0) | 12 | NA — No isolates of Streptococcus anginosus observed at baseline.
  Escherichia coli (19, 8) | 18 | 6
  Bacteroides fragilis (11, 1) | 10 | 1

6. Secondary Outcome: Number of Participants With Favorable Per-pathogen Microbiological Outcome Rate at Test Of Cure (TOC) Visit
Description: as for outcome 5
Time Frame: TOC (7 to 14 days after the last dose of study medication therapy)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Doripenem | Meropenem
Number analyzed (Participants) | 23 | 8
participants
  Streptococcus anginosus (13, 0) | 9 | NA — No isolates of Streptococcus anginosus observed at baseline.
  Escherichia coli (19, 8) | 15 | 5
  Bacteroides fragilis (11, 1) | 9 | 1

7. Secondary Outcome: Number of Participants With Favorable Per-pathogen Microbiological Outcome Rate at Late Follow-Up (LFU) Visit
Description: A total of 24 pathogens in the doripenem group and 6 pathogens in the meropenem group were isolated at baseline from the intra-abdominal culture and were susceptible to the study drug received. The most common pathogens isolated at baseline from the intra-abdominal culture are listed in the table below; the numbers in parenthesis next to each pathogen represent the number of participants with the pathogen isolated in the doripenem and meropenem treatment groups, respectively. The favorable per-pathogen microbiological outcome was considered when all baseline pathogens were eradicated (absence) or presumed eradicated (absence of material to culture in a participant who has a positive clinical response to treatment).
Time Frame: LFU (28 to 42 days after the last dose of study medication therapy)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Doripenem | Meropenem
Number analyzed (Participants) | 23 | 8
participants
  Streptococcus anginosus (13, 0) | 9 | NA — No isolates of Streptococcus anginosus observed at baseline.
  Escherichia coli (19, 8) | 15 | 5
  Bacteroides fragilis (11, 1) | 9 | 1

ADVERSE EVENTS:
Time Frame: Approximately 8 weeks
Arm/Group | Doripenem | Meropenem
Serious Adverse Events (participants affected / at risk) | 7/31 | 0/10
Other Adverse Events (participants affected / at risk) | 15/31 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doripenem (N=31) | Meropenem (N=10)
Abdominal Pain (Gastrointestinal disorders) | 3 | 0
Functional Gastrointestinal Disorder (Gastrointestinal disorders) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Abdominal Abscess (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Doripenem (N=31) | Meropenem (N=10)
Nausea (Gastrointestinal disorders) | 3 | 0
Abdominal Distension (Gastrointestinal disorders) | 2 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Tongue Ulceration (Gastrointestinal disorders) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 2 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 2 | 0
Electrocardiogram QT Prolonged (Investigations) | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 2 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Otitis Media (Infections and infestations) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated early due to business reasons and not related to safety concerns or issues. As such, the limited enrollment precludes a meaningful conclusion about the efficacy and safety of doripenem compared with meropenem.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days